CLINICAL TRIAL: NCT07138053
Title: The Impact of Multimodal Balancing Anesthesia vs Opioid Free Anesthesia on Postoperative Pain Intensity and Stress Response After Open Gynecology Surgery
Brief Title: The Impact Opioid Free Anesthesia on Postoperative Pain Intensity and Stress Response After Open Gynecology Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital Zenica (Other)
Responsible Party: Principal Investigator, Asmira Ljuca, MD Anesthesiologist and Intensive Care Subspecialist, Cantonal Hospital Zenica
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALJ07/25
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Opioid Free Anesthesia; Stress Response; Postoperative Pain
Keywords: opioid; cortisol; stress response
MeSH Terms: conditions — Fractures, Stress; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The diagnostic protocol was performed in patients at the gynecology department. The patients with diagnosed non cancer pathology and who needed gynecolog surgery were prepared for the surgical procedure. After that, patients were examined to a preoperative anesthetic visit. During the visit, participants were assessed according to eligibility for enrollment in the study. The participants who have met the eligibility criteria have explained the nature of the study protocol. Those who agreed to participate in the study were randomized to one of two study groups for the duration of the study.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Surgeons and outcome assessors were masking to the treatment allocation. Masking was impossible for anesthetist because anesthetist was performed different tip of anesthesia during surgery.
  The outcome study were evaluated by independent assessors who were also masked because they evaluated patients after surgery on a daily base during hospital stay without knowledge of the type intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MBA group (No Intervention): anesthesia based on opioids (multimodal balancing anesthesia with opioids)
- OFA group (Experimental): Experimental group will not receive opioids in perioperativ period
  Interventions: Other: OFA group

INTERVENTIONS:
Other: OFA group — OFA group Premedication with Midazolame and Paracetamol 30 minutes before surgery on ward, Dexamethasona and infusion of Dexmedetomidin and 2% Lidocaine 10 min before intubation( 50mcg Dexmedetomidin and 500mg 2% Lidocaine add up to 50ml normal saline) 1ml/10kg in 10 min after intubation 1ml/10kg/h discontinued after last surgical sutures. TAP bloc ultrasound guided performed after intubation. Ketamine given 60 sec before incision in doses 0.5 mg/kg, and after if it is necessary according to ER and qNOX. Provided value range between 40-60 during surgery.
  Arms: OFA group

SUMMARY:
This studi compared impact of multimodal balancing anesthesia vs opioid free anesthesia on postoperative pain intensity and stress response after open gynecology surgery.

Hypothesis was: opioid free anesthesia reduces postoperative pain intensity and stress response in terms of the value for pain in VAS (Visual Analog Scala) and for stress response in value of cortisol, prolactin and IL-6, CRP and improves postoperative patients subjective well-being and surgical outcome.

DETAILED DESCRIPTION:
This prospective randomized, controlled clinical study was carried out in the Department of Anesthesiology and Intensive Care Unit and Department of Gynecology at the Cantonal Hospital Zenica, Bosnia and Herzegovina. After obtaining ethical committee approval 80 participants, scheduled for elective open gynecology surgery were included into study. Sample size was estimated using sample size calculator software and power analysis with 90% confidence interval and power of 80%. Statistical significance was considered as p< 0,05. The calculation indicated 35 participants per group would be sufficient to detect a 50% difference for IL-6, cortisol, prolactin and CRP between the groups. Assuming dropout would lead to a total sample size of 80 participants. Before each participant agreed to the join the study, the purpose and procedures of the study were fully explained and informed and written consent was obtained from each participant. A preoperative anesthetic examination was conducted the day before surgery. The interventional group, opioid free anesthesia group(OFA group) and the control group, multimodal balancing anesthesia group (MBA group). Randomization was performed by computer generated randomization codes. The codes which indicated the treatment were held in sealed opaque envelopes. Nurse who conducted randomization and opened the envelopes the night before surgery was blinded to the study protocol as well as the gynecologist, nurses and staff involved in data collection.

The participants of MBA group were undergone to the traditional concept of preoperative and intraoperative anesthesia management with opioid. The participants in the intervention group received opioid free anesthesia and didn't received opioid in peroperativ period. Assessment of clinical parameters started at 06:00 am on the day of surgery (basal value). Peripheral venous blood samples were collected to measure serum levels of glucose, cortisol, prolactin, C-reactive protein, blood count and differential blood count and IL-6, and 06.00 am on the first postoperative day. Six hours post-surgery peripheral venous blood samples were collected to measure serum levels of glucose, cortisol, prolactin, blood count and differential blood count. All patients underwent to opioid free anesthesia will be given TAP block ultrasound guided after intubation and before surgical incision. Consciousness and pain respond monitored by Entropy or CONX device. Analgesia for opioid free arm during surgery will bi provided with combination of medicament (Dexmedetomidine, Ketamine, 2%Lidocaine, Dexamethasone and Magnesium sulfate). Blood pressure and hart rate recorded : before intubation, on intubation, skin incision, before extubation and two hour after extubation.

Assessment of subjective well-being was performed using a 10 cm horizontal Visual Analogue Scales for 1, 2, 4, 6-12 and 12-24 hours post-surgery. Pain at rest, pain with mobilization, thirst, hunger, mouth dryness, anxiety and weakness were evaluated. The patients were explained how to use the scale. Postoperative data included and the time to oral intake. The following data were recorded also: age, sex, body weight, body mass index, American Society of Anesthesiologists (ASA) physical status class, type of surgery.

ELIGIBILITY:
Inclusion Criteria:• participants with ASA physical status class I-II

* aged between 18 years and 65 years
* participants scheduled for elective open gynecology surgery non cancer

Exclusion Criteria:

body mass index above 30 kg/m2, diabetes mellitus, emergence surgery, cardiopulmonary disease, neuromusular disease, renal disease, vaginal hysterectomy, hepatic or endocrine disease, pregnancy, mental disease, allergy to any study drugs, alcoholic or drug abuse, ASA III and IV, patient's refusal to participate in the study, duration of surgery below 30min and over 90min.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-07-17 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative stress respons | blood samples were taken at 06:00am on the day of surgeon(basal value), 6 hours post-surgeon, at 06:00 am on the first postoperative day
  Primari mean in difference of strens respons beatween two group of patient meserments with value of cortisol, prolacti, IL-6 and C-reactive protein and glucosa blood level

SECONDARY OUTCOMES:
well-being score | The assessment of subjective well-being and pain score was performed 1,3,,6,12 ,24 and 48hours post-surgery]
  The mean change from baseline in participant's subjective well-being score on Visual Analogue Scale The participant's subjective well-being included: pain at rest and with movement, thirst, hunger, dry mouth, weakness, anxiety, nausea and vomiting. The mean change were measured using a 10 cm horizontal Visual Analogue Scale. The left end represented "no symptom" (score:0) and the right end represented "the worst imaginable" (score 10) limits of the variable to be evaluated. the scales line from score 0 to the patient's mark determined the score of symptom intensity.The score was calculated as follow: 0-1cm no symptom; 1-3 cm mild symptom; 3-7 cm moderate symptom; 7-10 cm strong symptom. The patients were questioned about presence of nausea and vomiting at six study time points. A "NO" answer was grade as 0 and a "YES" answer was graded as 1.

CONTACTS AND LOCATIONS:
Overall Officials: Asmira Ljuca, MD, Principal Investigator — Cantonal Hospital Zenica
Locations (1):
- Cantonal Hospital Zenica, Zenica, Zenica, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xia M, Ji NN, Duan ML, Tong JH, Xu JG, Zhang YM, Wang SH. Dexmedetomidine regulate the malignancy of breast cancer cells by activating alpha2-adrenoceptor/ERK signaling pathway. Eur Rev Med Pharmacol Sci. 2016 Aug;20(16):3500-6. PMID 27608913
- [Background] Lersch F, Correia PC, Hight D, Kaiser HA, Berger-Estilita J. The nuts and bolts of multimodal anaesthesia in the 21st century: a primer for clinicians. Curr Opin Anaesthesiol. 2023 Dec 1;36(6):666-675. doi: 10.1097/ACO.0000000000001308. Epub 2023 Sep 19. PMID 37724595
- [Background] Jameson P, Desborough JP, Bryant AE, Hall GM. The effect of cortisol suppression on interleukin-6 and white blood cell responses to surgery. Acta Anaesthesiol Scand. 1997 Feb;41(2):304-8. doi: 10.1111/j.1399-6576.1997.tb04683.x. PMID 9062617
- [Background] Helander EM, Webb MP, Bias M, Whang EE, Kaye AD, Urman RD. A Comparison of Multimodal Analgesic Approaches in Institutional Enhanced Recovery After Surgery Protocols for Colorectal Surgery: Pharmacological Agents. J Laparoendosc Adv Surg Tech A. 2017 Sep;27(9):903-908. doi: 10.1089/lap.2017.0338. Epub 2017 Jul 25. PMID 28742427
- [Background] Anand S, Bhati G, Gurram R, Gnanasekaran S, Kate V, Pottakkat B, Kalayarasan R. Does Neutrophil-to-Lymphocyte Ratio (NLR) Predict Pathologic Response to Neoadjuvant Chemoradiotherapy in Patients with Esophageal Squamous Cell Carcinoma? J Gastrointest Cancer. 2021 Jun;52(2):659-665. doi: 10.1007/s12029-020-00445-5. PMID 32607960
- [Background] Akeju O, Song AH, Hamilos AE, Pavone KJ, Flores FJ, Brown EN, Purdon PL. Electroencephalogram signatures of ketamine anesthesia-induced unconsciousness. Clin Neurophysiol. 2016 Jun;127(6):2414-22. doi: 10.1016/j.clinph.2016.03.005. Epub 2016 Mar 16. PMID 27178861
- [Background] Akeju O, Hobbs LE, Gao L, Burns SM, Pavone KJ, Plummer GS, Walsh EC, Houle TT, Kim SE, Bianchi MT, Ellenbogen JM, Brown EN. Dexmedetomidine promotes biomimetic non-rapid eye movement stage 3 sleep in humans: A pilot study. Clin Neurophysiol. 2018 Jan;129(1):69-78. doi: 10.1016/j.clinph.2017.10.005. Epub 2017 Oct 20. PMID 29154132